CLINICAL TRIAL: NCT06532136
Title: Treatment of Moderate-to-severe Papulopustular Rosacea With Deucravacitinib
Brief Title: Deucravacitinib Rosacea
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study is being closed due to sponsor withdrawal of funding and support.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Benjamin Ungar, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY-24-00593
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Papulopustular Rosacea
MeSH Terms: conditions — Rosacea | interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deucravacitinib (Active Comparator): Participants receiving 6mg deucravacitinib once daily for 8 weeks. Participants previously randomized to deucravacitinib will continue to receive deucravacitinib for an additional 8 weeks until Week 16.
  Interventions: Drug: Deucravacitinib
- Placebo then Deucravacitinib (Active Comparator): Participants receiving placebo once daily for 8 weeks. At week 8, those participants originally randomized to placebo will initiate dosing with 6mg deucravacitinib once daily for 8 weeks until Week 16.
  Interventions: Drug: Deucravacitinib; Drug: Placebo

INTERVENTIONS:
Drug: Deucravacitinib — Deucravacitinib 6 mg orally once daily.
Drug: Placebo — Matching placebo orally once daily.
  Arms: Placebo then Deucravacitinib

SUMMARY:
This will be a double-blind, randomized placebo-controlled study in which participants will be randomized 2:1 to receive 6 mg deucravacitinib or placebo once daily for 8 weeks, followed by an open label extension during which all participants will receive 6 mg deucravacitinib once daily for an additional 8 weeks. The open-label extension has been incorporated in order to ensure all participants receive benefit from the study, as well as to benefit from the intra-patient comparison of placebo to drug, and to provide longer-term clinical data.

The study will include 33 adult participants with moderate-to-severe Papulopustular Rosacea (PPR). participants will have baseline Investigator Global Assessment (IGA) score of at least 3 and at least 12 inflammatory lesions.

Beginning at Baseline/Week 0 enrolled participants will receive 6mg deucravacitinib or placebo once daily for 8 weeks. At week 8, those participants originally randomized to placebo will initiate dosing with 6mg deucravacitinib once daily for 8 weeks until Week 16. Participants previously randomized to deucravacitinib will continue to receive deucravacitinib for an additional 8 weeks until Week 16. All participants will return for visits at Weeks 4, 8, 12 and 16 following study treatment initiation for repeat clinical assessments, medication reviews, tape-strip collection, blood and urine sample collections, and monitoring for adverse events.

DETAILED DESCRIPTION:
After providing consent, all subjects will be assessed for study eligibility, which includes a review of the subjects past and current medical conditions, familial medical history and detailed review of past and current medications. Subjects will also undergo a review of past topical treatments/therapies for PPR, and clinical assessments (inflammatory lesion count, IGA, CEA, PSA). Subjects will have urine (for urinalysis) and blood (for Complete Blood Count with differential, Comprehensive Metabolic Panel, lipid panel, creatinine kinase, C-Reactive Protein, HIV, HCV and HBV) collected for safety analysis. In addition, subjects will be screened for tuberculosis via PPD or quantiferon gold testing, and pregnancy (if applicable) via serum pregnancy test.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥ 18 years of age at the time of signing the informed consent document.
* Participant is able to understand and voluntarily sign an informed consent document prior to participation in any study assessments or procedures.
* Participant is able to adhere to the study visit schedule and other protocol requirements.
* Diagnosis of PPR, baseline IGA ≥ 3, and baseline inflammatory lesion count ≥ 12
* Participant agrees to discontinue all treatments for PPR from screening through study completion aside from the study drug
* Participant is judged to be in otherwise good overall health as judged by the investigator, based on medical history, physical examination, and laboratory testing. (NOTE: The definition of good health means a participant does not have uncontrolled significant co-morbid conditions).
* Participant agrees not to receive a live vaccine during the study and for at least 4 weeks after the last study drug dose.
* Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. While on the study drug and for at least 90 days after the last dose of the study drug, male and female participants must be willing to take appropriate contraceptive measures to avoid pregnancy or fathering a child. FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

  * Option 1: Any one of the following highly effective contraceptive methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy OR
  * Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]); PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

The female participant's chosen form of contraception must be effective by the time the female participant is enrolled into the study.

Exclusion Criteria:

The presence of any of the following will exclude a participant from enrollment:

* Participants with other skin diseases that would interfere with the study assessment in the opinion of the investigator.
* Active bacterial, fungal, or viral skin infection within 2 weeks from study initiation.
* Participants has clinically significant (as determined by the investigator) renal, hepatic, hematologic, intestinal, endocrine, pulmonary, cardiovascular, neurological, psychiatric, immunologic, or other major uncontrolled diseases (e.g., malignancy, TB, HIV, HBV, HCV, thromboembolic events) that will affect the health of the participant during the study or interfere with the interpretation of study results.
* Participant has previously received treatment with TYK2 inhibitor
* Current topical or oral treatments (e.g., topical corticosteroids, topical calcineurin inhibitors, topical JAK inhibitors, topical metronidazole, topical minocycline, topical ivermectin, topical azelaic acid, topical brimonidine, topical oxymetazoline oral antibiotics) within 2 weeks of baseline
* Use of systemic immunosuppressive medications, including, but not limited to, cyclosporine, systemic or intralesional corticosteroids, mycophenolate mofetil, azathioprine, methotrexate, tacrolimus within 4 weeks of study initiation
* History of adverse systemic or allergic reactions to any component of the study drug.
* Current participation in any other study with an investigational medication
* Participant who is pregnant or breast feeding or plans on becoming pregnant or breastfeeding
* Participant has received a live vaccine < 4 weeks of Baseline/Week 0 visit.
* ANY of the following abnormalities in the clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat, if deemed necessary

  * Absolute neutrophil count of <1.2 x 109/L (<1200/mm3);
  * Hemoglobin <11.0 g/dL or hematocrit <33%;
  * Platelet count of <150 x 109/L (<150,000/mm3);
  * Absolute lymphocyte count of <0.80 x 109 /L (<800/mm3);
  * Estimated Glomerular Filtration Rate (eGFR) less than 60 mL/ml/min/1.73m2 based on CKD-Epi 2021 (creatine equation);
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) values >2 times the ULN;
  * Total bilirubin ≥ 1.5 times the ULN; participants with a history of Gilbert's syndrome may have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin is ≤ ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Percent change in inflammatory lesion (papule/pustule) count | Baseline and Week 8
  This outcome looks at the percent change in inflammatory lesion presence (papule/pustule) from Baseline and Week 8 in deucravacitinib-treated vs. placebo patients. Lesions will be physically counted.

SECONDARY OUTCOMES:
Investigator Global Assessment (IGA) Success | Baseline, Week 4, Week 4, Week 8, Week 12, Week 16
  IGA Success is defined by a clear (0) or almost clear (1) and a reduction from baseline of ≥ 2 points score of 0 or 1 at weeks 4, 8, 12, and 16 in deucravacitinib-treated patients.
  IGA is a 5-point scale defined by the following parameters: 0 (clear), 1 (almost clear), 2 (mild disease), 3 (moderate disease), 4 (severe disease), with higher rating indicating more severe outcomes.
The Clinical Erythema Assessment | Week 4, Week 4, Week 8, Week 12, Week 16
  The Clinical Erythema Assessment assesses the redness of skin. This outcome is measuring change in erythema.
  It is defined by the following parameters: 0 - Clear (clear skin with no signs of erythema), 1 - Almost Clear (almost clear, slight redness), 2 - Mild (mild erythema; definite redness), 3 - Moderate (moderate erythema; marked redness), 4 - Severe (severe erythema; fiery redness). Higher rating indicates more severe outcomes.
The Clinical Patient Severity Assessment | Baseline, Week 4, Week 4, Week 8, Week 12, Week 16
  The Clinical Patient Severity Assessment assesses the patient's perspective of the redness of their skin. This outcome is measuring change in patient's perspective of erythema.
  It is defined by the following parameters: 0 - Clear (clear of unwanted redness), 1 - Almost Clear (nearly clear of wanted redness), 2 - Mild (somewhat more redness than I prefer), 3 - Moderate (more redness than I prefer), 4 - Severe (completely unacceptable redness).
Change from baseline in The Dermatology Life Quality Index (DLQI | Baseline, Week 4, Week 4, Week 8, Week 12, Week 16
  The Dermatology Life Quality Index (DLQI) measures how much the patient's rosacea has affected their life over the previous week. It is a 10 question instrument. This outcome is measuring change in quality of life impaired by rosacea.
  The answer to each question is scored according to the following: Question unanswered - scored 0, Not relevant - scored 0, Not at all - scored 0, A little - scored 1, A lot - scored 2, Very much - scored 3. The DLQI is calculated by summing the score of each question. The maximum score is 30 and the minimum score is 0. A higher score represents a quality of life that is more impaired. Overall DLQI scores are defined as 0-1 = no effect at all on patient's life, 2-5 = small effect on patient's life, 6-10 = moderate effect on patient's life, 11 - 20 = very large effect on patient's life, 21 -30 = extremely large effect on patient's life.
Change from baseline in Ocular Surface Disease Index (OSDI) | Baseline, Week 4, Week 4, Week 8, Week 12, Week 16
  The Ocular Surface Disease Index (OSDI) is used for measuring dry eye disease in patients. This outcome is measuring change in dry eye disease and effect on vision-related function.
  OSDI is a 12 question instrument. The answer to each question is scored according to the following: All of the time - scored 4, Most of the time - scored 3, Half of the time - scored 2, Some of the time - scored 1, None of the time - scored 0. OSDI is assessed on a scale of 0 to 100, with higher scores representing greater disability.
Change in Inflammatory (papule/pustule) lesion count | Baseline, Week 8, Week 16
  Change from Baseline and from Week 8 in inflammatory (papule/pustule) lesion count at Week 16. A lesser lesion count at Week 16 indicates disease improvement.
Change from baseline in IGA score at 4, 8, 12, and 16 weeks | Baseline, Week 4, Week 4, Week 8, Week 12, Week 16
  Change from Baseline in IGA score at Week 4, 8, 12, and 16.
  IGA is a 5-point scale defined by the following parameters: 0 (clear), 1 (almost clear), 2 (mild disease), 3 (moderate disease), 4 (severe disease). A decrease in IGA indicated improvement in disease, while an increase in IGA indicates worsening disease.
Percent change from baseline in IGA score at 4, 8, 12, and 16 weeks | Baseline, Week 4, Week 4, Week 8, Week 12, Week 16
  Percent change from Baseline in IGA score at Week 4, 8, 12, and 16.
  IGA is a 5-point scale defined by the following parameters: 0 (clear), 1 (almost clear), 2 (mild disease), 3 (moderate disease), 4 (severe disease). A decrease in IGA indicated improvement in disease, while an increase in IGA indicates worsening disease.
Frequency Adverse Events (AEs) | Baseline, Week 4, Week 4, Week 8, Week 12, Week 16
  Safety and tolerability will be evaluated from the frequency of AEs.
Duration of AEs | Baseline, Week 4, Week 4, Week 8, Week 12, Week 16
  Safety and tolerability will be evaluated from the duration of AEs. This outcome will assess the safety of treatment.
Severity of AEs | Baseline, Week 4, Week 4, Week 8, Week 12, Week 16
  Safety and tolerability will be evaluated from the severity of AEs.
  Severity of AEs is measured through a grading system Common Terminology Criteria for Adverse Events (CTCAE), which assigns severity grades ranging from 1 to 5. The scale is as follows:
  Grade 1: Mild Grade 2: Moderate Grade 3: Severe Grade 4: Potentially life-threatening Grade 5: Results in Death Mild is defined as not significantly interfering with the patient's usual function. Moderate is defined as interfering to some extent with the patient's usual function. Severe is defined as preventing the patient from performing their usual functions.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Ungar, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Results will be provided as aggregated data.